CLINICAL TRIAL: NCT01078662
Title: A Phase II, Open Label, Non Randomised, Non Comparative, Multicentre Study to Assess the Efficacy and Safety of Olaparib Given Orally Twice Daily in Patients With Advanced Cancers Who Have a Confirmed Genetic BRCA 1 and/or BRCA2 Mutation
Brief Title: Open Label Study to Assess Efficacy and Safety of Olaparib in Confirmed Genetic BRCA1 or BRCA2 Mutation Pats
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00042; 2010-022278-15 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Ovarian; Breast; Prostate; Pancreatic; Advanced Tumours
Keywords: olaparib; PARP inhibitors; genetic BRCA1 mutation; BRCA2 mutation; solid tumour refractory
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Olaparib is available as a film-coated tablet containing 150 mg or 100 mg of olaparib. Subjects will be administered study treatment orally at a dose recommended by Investigator. Full dose: 300 mg twice daily (bid) or Reduced doses: 200 mg twice daily (bid) or 100 mg twice daily (bid). The planned dose of 300 mg bid will be made up of two x 150 mg tablets twice daily, with 100 mg tablets used to manage dose reductions.
  Interventions: Drug: olaparib

INTERVENTIONS:
Drug: olaparib — Tablets Oral BID
  Other Names: Lynparza

SUMMARY:
To assess the efficacy of oral olaparib in patients with advanced cancer who have a confirmed genetic BRCA1 and/or BRCA2 mutation, by assessment of tumour response

ELIGIBILITY:
Inclusion Criteria:

* Confirmed documented deleterious or suspected deleterious BRCA mutation. (The presence of a loss-of-function germline mutation in the BRCA1 and/or BRCA2 gene must be confirmed prior to consent according to local practice).
* Confirmed malignant solid tumours for which no standard treatment exists
* At least one lesion (measurable and/or non measurable) at baseline that can be accurately assessed by CT/MRI and is suitable for repeated assessment at follow up visits

Exclusion Criteria:

* Any previous treatment with a PARP inhibitor, including olaparib
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Patients receiving any systematic chemotherapy, radiotherapy (except for palliative reasons) within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2010-02-21 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Bella Kaufman, MD, Principal Investigator — Chaim Sheba Medical Centre, Tel Hashomer, Israel
Locations (12):
- United States (2):
  - Research Site, West Hollywood, California
  - Research Site, Philadelphia, Pennsylvania
- Australia (2):
  - Research Site, Melbourne
  - Research Site, Randwick
- Research Site, Cologne, Germany
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Research Site, Madrid, Spain
- Research Site, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Matulonis UA, Penson RT, Domchek SM, Kaufman B, Shapira-Frommer R, Audeh MW, Kaye S, Molife LR, Gelmon KA, Robertson JD, Mann H, Ho TW, Coleman RL. Olaparib monotherapy in patients with advanced relapsed ovarian cancer and a germline BRCA1/2 mutation: a multistudy analysis of response rates and safety. Ann Oncol. 2016 Jun;27(6):1013-1019. doi: 10.1093/annonc/mdw133. Epub 2016 Mar 8. PMID 26961146
- [Derived] Domchek SM, Aghajanian C, Shapira-Frommer R, Schmutzler RK, Audeh MW, Friedlander M, Balmana J, Mitchell G, Fried G, Stemmer SM, Hubert A, Rosengarten O, Loman N, Robertson JD, Mann H, Kaufman B. Efficacy and safety of olaparib monotherapy in germline BRCA1/2 mutation carriers with advanced ovarian cancer and three or more lines of prior therapy. Gynecol Oncol. 2016 Feb;140(2):199-203. doi: 10.1016/j.ygyno.2015.12.020. Epub 2015 Dec 23. PMID 26723501
- See also: Protocol redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1678&filename=D0810C00042_Clinical_Study_Protocol_redacted_[SECURED].pdf
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0810C00042&attachmentIdentifier=b8b9546d-a241-4531-b6eb-f5ad8d2ee85b&fileName=Clinical_Study_Protocol_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 sites across Israel, Germany, Spain, Australia, USA, Sweden. Enrolment started in Feb 2010 and was completed in Jul 2012. In total, 298 patients had received treatment (olaparib).
Pre-assignment Details: Patients >17 years age with histologically and/or cytologically confirmed malignant solid tumours, refractory to standard therapy for which no suitable effective/curative therapy. Patients with confirmed deleterious or suspected deleterious BRCA mutation, Eastern Co-operative Oncology Group performance status ≤2 and life expectancy of ≥12 weeks.
  In total, 298 patients had received treatment.
Groups:
- Breast Cancer: Patients with primary cancer site = breast. Receiving olaparib 400mg BID
- Ovarian Cancer: Patients with primary cancer site = ovary. Receiving olaparib 400mg BID
- Pancreatic Cancer: Patients with primary cancer site = pancreas. Receiving olaparib 400mg BID
- Prostate Cancer: Patients with primary cancer site = prostate. Receiving olaparib 400mg BID
- Other Cancers: Patients with other primary cancers. Receiving olaparib 400mg BID
Period: Overall Study
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer | Other Cancers
Started | 62 | 193 | 23 | 8 | 12
Completed | 4 | 25 | 2 | 1 | 1
Not Completed | 58 | 168 | 21 | 7 | 11
Not completed — Death | 41 | 103 | 18 | 5 | 8
Not completed — Patients reached data cut-off | 12 | 53 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 4 | 11 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer | Other Cancers | Total
Number analyzed (Participants) | 62 | 193 | 23 | 8 | 12 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of screening
  years | 47.6 (9.69) | 57.2 (9.28) | 57.1 (7.99) | 66.6 (9.86) | 54.9 (12.38) | 55.3 (10.3)
Age, Customized [Count of Participants; unit: Participants] — Age by category
  Participants
    < 50 years | 33 | 40 | 6 | 0 | 4 | 83
    >=50 to <65 years | 28 | 117 | 14 | 3 | 5 | 167
    >= 65 years | 1 | 36 | 3 | 5 | 3 | 48
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 61 | 193 | 10 | 0 | 8 | 272
    Male | 1 | 0 | 13 | 8 | 4 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 60 | 183 | 21 | 8 | 11 | 283
    Black or African American | 0 | 1 | 1 | 0 | 0 | 2
    Asian | 1 | 8 | 1 | 0 | 1 | 11
    Other | 1 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumour Response Rate
Description: Tumour response rate is the proportion of patients who experienced complete or partial response at least once during the assessment period, according to the definitions of Response Evaluation Criteria In Solid Tumours (RECIST version 1.1).
Time Frame: Tumour assessments carried out at baseline ie 28 days before first study drug dose and then every 8 weeks up to 6 months after starting study treatment, then every 12 weeks until objective disease progression, assessed maximum up to 29 months
Population: Full analysis set - all treated patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Patients: Patients of different cancer types
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer | Other Cancers | All Patients
Number analyzed (Participants) | 62 | 193 | 23 | 8 | 12 | 298
Percentage of participants | 12.9 [5.74 to 23.85] | 31.1 [24.64 to 38.13] | 21.7 [7.46 to 43.7] | 50 [15.7 to 84.3] | 8.3 [0.21 to 38.48] | 26.2 [21.27 to 31.55]

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate is the proportion of patients with at least one measurable lesion at baseline, who experienced complete or partial response at least once during the assessment period, according to the definitions of Response Evaluation Criteria In Solid Tumours (RECIST version 1.1).
Time Frame: as for outcome 1
Population: Measurable disease analysis set - all treated patients having at least one measurable lesion at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer | Other Cancers | All Patients
Number analyzed (Participants) | 58 | 167 | 23 | 7 | 11 | 266
Percentage of participants | 13.8 [6.15 to 25.38] | 35.9 [28.66 to 43.7] | 21.7 [7.46 to 43.7] | 57.1 [18.41 to 90.1] | 9.1 [0.23 to 41.28] | 29.3 [23.92 to 35.19]

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the duration from first dose till objective progression or death. In absence of progression or death, the time is calculated from first dose till last evaluable scanning visit.
Time Frame: Tumour assessments are carried out at baseline ie 28 days before first study drug dose and then every 8 weeks up to 6 months after starting study treatment, then every 12 weeks until objective disease progression, assessed maximum up to 29 months
Population: Full analysis set - all treated patients. The Other cancer group was not analysed in accordance with the protocol.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer
Number analyzed (Participants) | 62 | 193 | 23 | 8
months | 3.68 [1.76 to 7.52] | 7.03 [3.65 to 11.24] | 4.55 [1.81 to 8.21] | 7.15 [2.63 to 17.45]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration from first dose till death. In absence of death, the time is calculated from first dose till the date subject last known to be alive.
Time Frame: Survival follow-up from first dose till death of the patient or till end of study in absence of death, assessed maximum up to 29 months
Population: Full analysis set - all treated patients. The Other cancer group was not analysed in accordance with the protocol.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer
Number analyzed (Participants) | 62 | 193 | 23 | 8
months | 11.01 [5.68 to 24.18] | 16.62 [9.43 to NA] — No enough data to calculate upper limit | 9.81 [3.84 to 16.62] | 18.38 [6.24 to 25.46]

5. Secondary Outcome: Overall Survival Rate at 12 Months
Description: Overall survival rate at 12 months is defined as the proportion of patients who are alive 12 months after date of first dose
Time Frame: as for outcome 4
Population: Full analysis set - all treated patients. The Other cancer group was not analysed in accordance with the protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer
Number analyzed (Participants) | 62 | 193 | 23 | 8
Percentage of participants | 44.7 [5.68 to 24.18] | 64.4 [9.43 to NA] | 40.9 [3.84 to 16.62] | 50 [6.24 to 25.46]

6. Secondary Outcome: Duration of Response
Description: Duration of response is calculated from the date of first documented response (complete or partial) until date of documented progression (as defined by RECIST 1.1) or death (by any cause) in the absence of disease progression.
Time Frame: From onset of first occurrence of complete or partial response till documented progression or death by any cause in the absence of progression, assessed maximum up to 29 months
Population: Full analysis set - all treated patients who had at least one complete or partial response during the assessment period.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer | Other Cancers | All Patients
Number analyzed (Participants) | 8 | 60 | 5 | 4 | 1 | 78
days | 204 [149.5 to 405] | 225 [143 to 410] | 134 [131 to 141] | 326.5 [164 to 476] | 165 [165 to 165] | 208 [134 to 410]

7. Secondary Outcome: Disease Control Rate at Week 16
Description: Disease control rate is the proportion of patients with best response of complete or partial response or stable disease according to definitions of Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) till week 16.
Time Frame: Tumour assessments carried out at baseline ie 28 days before first study drug dose and then at week 8 and week 16
Population: Full analysis set - all treated patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Breast Cancer | Ovarian Cancer | Pancreatic Cancer | Prostate Cancer | Other Cancers | All Patients
Number analyzed (Participants) | 62 | 193 | 23 | 8 | 12 | 298
Percentage of participants | 37.1 [25.16 to 50.31] | 58 [50.73 to 65.08] | 47.8 [26.82 to 69.41] | 62.5 [24.49 to 91.48] | 33.3 [9.92 to 65.11] | 52 [46.18 to 57.81]

ADVERSE EVENTS:
Arm/Group | OLAPARIB
Serious Adverse Events (participants affected / at risk) | 90/298
Other Adverse Events (participants affected / at risk) | 290/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLAPARIB (N=298)
ANAEMIA (Blood and lymphatic system disorders) | 13 (14)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3)
ENTERITIS (Gastrointestinal disorders) | 1 (1)
INTESTINAL MASS (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 7 (8)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (3)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
DIPLOPIA (Eye disorders) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (12)
ASCITES (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 3 (4)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 7 (9)
VOMITING (Gastrointestinal disorders) | 5 (6)
DEVICE OCCLUSION (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 3 (3)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
ENTEROBACTER SEPSIS (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 4 (4)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (2)
SEPSIS (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (3)
SYNCOPE (Nervous system disorders) | 2 (2)
ANXIETY (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLAPARIB (N=298)
ANAEMIA (Blood and lymphatic system disorders) | 90 (120)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 28 (36)
DRY MOUTH (Gastrointestinal disorders) | 19 (20)
DYSPEPSIA (Gastrointestinal disorders) | 52 (54)
ASTHENIA (General disorders) | 25 (33)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 17 (18)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 16 (18)
LEUKOPENIA (Blood and lymphatic system disorders) | 23 (35)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 33 (35)
ABDOMINAL PAIN (Gastrointestinal disorders) | 66 (85)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 25 (27)
CONSTIPATION (Gastrointestinal disorders) | 42 (53)
DIARRHOEA (Gastrointestinal disorders) | 81 (103)
FLATULENCE (Gastrointestinal disorders) | 23 (28)
NAUSEA (Gastrointestinal disorders) | 176 (218)
VOMITING (Gastrointestinal disorders) | 109 (158)
FATIGUE (General disorders) | 176 (199)
OEDEMA PERIPHERAL (General disorders) | 41 (48)
PYREXIA (General disorders) | 37 (51)
NASOPHARYNGITIS (Infections and infestations) | 23 (26)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 23 (29)
URINARY TRACT INFECTION (Infections and infestations) | 30 (44)
BLOOD CREATININE INCREASED (Investigations) | 21 (21)
WEIGHT DECREASED (Investigations) | 26 (26)
DECREASED APPETITE (Metabolism and nutrition disorders) | 62 (67)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 (33)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 37 (43)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 27 (31)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 15 (16)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 25 (26)
DIZZINESS (Nervous system disorders) | 34 (34)
DYSGEUSIA (Nervous system disorders) | 47 (47)
HEADACHE (Nervous system disorders) | 48 (60)
ANXIETY (Psychiatric disorders) | 17 (17)
DEPRESSION (Psychiatric disorders) | 19 (19)
INSOMNIA (Psychiatric disorders) | 22 (22)
COUGH (Respiratory, thoracic and mediastinal disorders) | 42 (52)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 36 (44)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 15 (15)
RASH (Skin and subcutaneous tissue disorders) | 15 (16)
HOT FLUSH (Vascular disorders) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less